CLINICAL TRIAL: NCT01432353
Title: An Open-label, Multicenter, Phase I Trial of the Safety and Pharmacokinetics of Escalating Doses of DFRF4539A in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of DFRF4539A in Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRF4998g; GO27825 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-09-08; First posted 2011-09-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: DFRF4539A

INTERVENTIONS:
Drug: DFRF4539A — multiple ascending doses

SUMMARY:
This multicenter, open-label, dose-escalating study will assess the safety and efficacy of DFRF4539A in patients with relapsed or refractory multiple myeloma. Cohorts of patients will receive multiple ascending doses of intravenous DFRF4539A every 3 weeks or weekly. Patients exhibiting acceptable safety and evidence of clinical benefit may receive DFRF4539A for up to 17 cycles. Anticipated time on study treatment is 1 year or until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients; >/= 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Relapsed or refractory multiple myeloma for which no effective standard therapy exists
* One of the prior therapies must have included a proteosome inhibitor or an immunomodulatory drug
* Measurable disease as defined by protocol

Exclusion Criteria:

* Prior use of monoclonal antibody within 4 weeks before Cycle 1, Day 1
* Treatment with radiotherapy, thalidomide, lenalidomide, bortezomib, any chemotherapeutic agent, or treatment with any investigational anti-cancer agent within 2 weeks prior to Cycle 1, Day 1
* Toxicities from any previous treatment must be resolved prior to Cycle 1, Day 1, except for neuropathy
* Completion of autologous stem cell transplant within 100 days prior to Cycle 1, Day 1
* Prior allogeneic stem cell transplant
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Grade > 1 peripheral neuropathy
* Active infection at screening or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 4 weeks prior to Cycle 1, Day 1
* Positive for hepatitis B, hepatitis C or HIV infection
* Pregnant or lactating women or women who intend to become pregnant within the period of time of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 3.5 years
Safety: Maximum tolerated dose/dose-limiting toxicities | approximately 1.5 years
Recommended Phase II dose for every-3-week or weekly administration of DFRF4539A | approximately 3.5 years

SECONDARY OUTCOMES:
Immunogenicity: Serum antitherapeutic antibody levels | approximately 3.5 years
Pharmacokinetics: Area under the concentration - time curve (AUC) | approximately 3.5 years
Objective response, tumor assessments according to International Myeloma Working Group (IMWG) Uniform Response Criteria and/or European Bone Marrow Transplant (EBMT) Criteria | approximately 3.5 years
Duration of objective response, defined as time from first documented objective response to progression or death of any cause | approximately 3.5 years
Progression-free survival, defined as time from first study treatment (Cycle 1, Day 1) to disease progression or death during study or within 30 days after last dose of study drug, whichever occurs first | approximately 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (8):
- United States (8):
  - Scottsdale, Arizona
  - Duarte, California
  - Jacksonville, Florida
  - Sarasota, Florida
  - Chicago, Illinois
  - Bethesda, Maryland
  - New York, New York
  - Nashville, Tennessee